CLINICAL TRIAL: NCT06133543
Title: RAISN - Robot-assisted ICG-guided Sentinel Node Biopsy in Testicular Cancer
Brief Title: Robot-assisted ICG-guided Sentinel Node Biopsy in Testicular Cancer
Acronym: RAISN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Intuitive Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2328
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Germ Cell Tumor; Seminoma; Nonseminomatous Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Seminoma; Nonseminomatous germ cell tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Negative sentinel lymph node (Experimental): Patients with negative sentinel lymph node biopsy are enrolled to active surveillance after surgery
  Interventions: Procedure: Robot-assisted ICG-guided sentinel lymph node biopsy
- Positive sentinel lymph node (Experimental): Patients with positive lymph node biopsy undergo a template retroperitoneal lymph node dissection in the same procedure
  Interventions: Procedure: Robot-assisted ICG-guided sentinel lymph node biopsy

INTERVENTIONS:
Procedure: Robot-assisted ICG-guided sentinel lymph node biopsy — The robot-assisted ICG-guided sentinel node (SN) biopsy is conducted as follows: At the start of the operation, indocyanine green (ICG) solution is transscrotally injected into the testicular parenchyma. The patient is positioned in the nephrectomy posture. After port placement and docking of the robotic system, the sentinel node(s) should be visible with the fluorescence camera. The SN is removed and sent for immediate frozen section biopsy evaluation. The inguinal orchiectomy is performed subsequently until the biopsy results are available. If the biopsy is negative, the procedure concludes. If the biopsy shows viable tumor, indicating clinical stage IIA and the indication for systematic unilateral retroperitoneal lymph node dissection. The patient was informed about the potential expansion of the procedure upon study enrollment. After the procedure, all patients are placed under observation and do not receive adjuvant systemic treatment. The follow-up period extends to 2 years.

SUMMARY:
Robot-assisted image-guided sentinel lymph node biopsy (RAISN) in testicular cancer is a novel technique that has not been widely investigated yet. This technique is promising and could be implemented as a future standard in the primary diagnostic work up of clinical stage (CS) I testicular cancer. Current staging strategies have a poor predictive accuracy for occult metastatic disease.

So far, feasibility studies used 99mTC-nanocolloid staining and laparoscopy and all patients with tumor-positive nodes received adjuvant systemic treatment. The development of a robot-assisted image-guided lymph node resection technique with indocyanine green (ICG) is potentially more precise, easier to apply and widely available. With this new diagnostic approach the management of newly diagnosed testicular cancer patients might be changed dramatically by reducing overtreatment and treatment-related toxicity with a minimally invasive robot-assisted procedure.

DETAILED DESCRIPTION:
The sentinel lymph node biopsy in testicular cancer is a novel technique that has not been extensively studied. This technique shows promise and could potentially become the future standard in the primary diagnosis of testicular cancer in clinical stage I.

In cases of clinical stage I testicular cancer, 20% to 30% of patients experience a recurrence. Strategies such as adjuvant chemotherapy or retroperitoneal lymph node dissection can reduce the risk of recurrence to 2% and 9%, respectively. However, the issue with these strategies is that the majority of patients may receive unnecessary treatment and endure the toxicity of chemotherapy or surgery. German and European guidelines recommend a risk-adapted approach. Testicular tumor patients with specific histopathological features are classified into low and high risk, with adjuvant therapy recommended accordingly. This strategy allows for more targeted treatment but still maintains a limited sensitivity of approximately 73%.

There have been few studies investigating the possibility of sentinel lymph node diagnostics in testicular cancer. Reasons for this include the rarity of the disease coupled with a lack of experience in minimally invasive surgery for testicular cancer treatment. Previous sentinel lymph node studies utilized the radioligand technique with technetium, which was limited to centers with a nuclear medicine department. With the advancing development of robotics and fluorescence technology using indocyanine green, there is an opportunity for a novel, minimally invasive lymph node diagnostic method applicable on a broader scale for testicular cancer patients.

In previous feasibility studies on sentinel lymph node diagnostics in testicular tumor patients, the use of 99mTC-nanocolloid staining and laparoscopy achieved a 90% sensitivity. The development of a robot-assisted image-guided lymph node resection technique using indocyanine green (ICG) is potentially more precise, easier to apply, and generally more available. Multiple studies in other tumor entities have demonstrated the non-inferiority and superiority of ICG over technetium. This new diagnostic approach could drastically change the treatment for newly diagnosed testicular cancer patients by reducing overtreatment and treatment-related toxicity through a minimally invasive robot-assisted procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed unequivocal testicular tumor by palpation and sonography with or without elevation of specific tumor markers AFP and/or ß-HCG.
* Clinical exclusion of metastases in preoperative staging using contrast-enhanced CT of the thorax and abdomen.
* The patient is of legal age.
* The patient can communicate with the investigator without issues or limitations and can understand and sign the patient information and consent form without problems or limitations.

Exclusion Criteria:

* Testicular tumor with uncertain dignity
* Patients with small testicular masses (< 1 cm)
* Patients with prior scrotal or retroperitoneal surgery for reasons other than a germ cell tumor.
* The patient has received different chemotherapy.
* The patient has undergone retroperitoneal radiotherapy.
* Exclusion criteria for the use of ICG include a history of anaphylactic reactions to ICG and iodine intolerance (ICG solution contains sodium iodide).
* The patient is in a reduced general condition or has a life-threatening illness.
* The patient has a psychiatric illness.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  The primary endpoint of the study is to demonstrate that RAISN has a sensitivity of ≥ 90% in nodal staging for testicular tumors in clinical stage I.

SECONDARY OUTCOMES:
Complications | 2 years
  EAUiaiC-classification and Clavien Dindo
Retrograde ejaculation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided